CLINICAL TRIAL: NCT01427179
Title: Genetic Investigations in Spontaneous Coronary Artery Dissection (SCAD)
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sharonne Hayes, Principal Investigator, Mayo Clinic
Other Study IDs: 11-000160
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Spontaneous Coronary Artery Dissection; SCAD
Keywords: Spontaneous coronary artery dissection; SCAD
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A 30 ml sample of blood from a vein or an existing catheter will be drawn at Mayo Clinic or another medical center and returned through the mail in a kit. Alternatively, a saliva sample will be collected and returned through the mail in a kit. An additional 10 ml (2 teaspoons) of blood, buccal smear, and/or available tissue samples may also be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the research is to identify mutations (defects in the genetic blueprint) that cause spontaneous coronary artery dissection (SCAD), in other words, spontaneous tears in blood vessels that supply the heart.

Some mutations may be inherited (passed on) from a parent without an apparent blood vessel problem while others may develop for the first time in the affected person.

DETAILED DESCRIPTION:
Study question: Do mutations within certain genes cause or confer susceptibility to spontaneous coronary artery dissection (SCAD)?

Specific aims:

1. Create a genomic DNA and plasma biobank for individuals diagnosed with SCAD.
2. Identify inherited and de novo/new mutations that underlie SCAD.
3. Identify common genetic variants that confer risk for SCAD.

Long term objective:Discover molecular and cellular mechanisms of SCAD and develop biomarkers to enable prediction and prevention.

The purpose of the research is to identify mutations (defects in the genetic blueprint) that cause tears in blood vessels that supply the heart. Some mutations may be inherited (passed on) from a parent without an apparent blood vessel problem while others may develop for the first time in the affected person. The study includes individuals diagnosed with spontaneous coronary artery dissection, their biological parents, and relatives with fibromuscular dysplasia, arterial aneurysm, or arterial dissection.

Adults with SCAD will be identified both retrospectively and prospectively.Confirmation of the diagnosis by review of coronary angiography will be required before proceeding with the informed consent process and blood or saliva sample procurement.

ELIGIBILITY:
Inclusion Criteria:

* Men and women able to give informed consent and complete a 2 page questionnaire
* Diagnosis of one or more episodes of spontaneous coronary artery dissection (SCAD)
* Biological parent of individual with SCAD
* Relative with fibromuscular dysplasia, arterial aneurysm, or arterial dissection

Exclusion Criteria:

* Lack of confirmation of SCAD diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with spontaneous coronary artery dissection (SCAD), their biological parents, and relatives with fibromuscular dysplasia, arterial aneurysm, or arterial dissection.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-05; Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of one or more gene mutation responsible for SCAD | By end of study
  Via GWAS and whole exome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sharonne N. Hayes, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tweet MS, Gulati R, Aase LA, Hayes SN. Spontaneous coronary artery dissection: a disease-specific, social networking community-initiated study. Mayo Clin Proc. 2011 Sep;86(9):845-50. doi: 10.4065/mcp.2011.0312. PMID 21878595
- [Background] Hayes SN, Kim ESH, Saw J, Adlam D, Arslanian-Engoren C, Economy KE, Ganesh SK, Gulati R, Lindsay ME, Mieres JH, Naderi S, Shah S, Thaler DE, Tweet MS, Wood MJ; American Heart Association Council on Peripheral Vascular Disease; Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Genomic and Precision Medicine; and Stroke Council. Spontaneous Coronary Artery Dissection: Current State of the Science: A Scientific Statement From the American Heart Association. Circulation. 2018 May 8;137(19):e523-e557. doi: 10.1161/CIR.0000000000000564. Epub 2018 Feb 22. PMID 29472380
- [Background] Goel K, Tweet M, Olson TM, Maleszewski JJ, Gulati R, Hayes SN. Familial spontaneous coronary artery dissection: evidence for genetic susceptibility. JAMA Intern Med. 2015 May;175(5):821-6. doi: 10.1001/jamainternmed.2014.8307. PMID 25798899
- [Background] Henkin S, Negrotto SM, Tweet MS, Kirmani S, Deyle DR, Gulati R, Olson TM, Hayes SN. Spontaneous coronary artery dissection and its association with heritable connective tissue disorders. Heart. 2016 Jun 1;102(11):876-81. doi: 10.1136/heartjnl-2015-308645. Epub 2016 Feb 10. PMID 26864667
- [Background] Adlam D, Olson TM, Combaret N, Kovacic JC, Iismaa SE, Al-Hussaini A, O'Byrne MM, Bouajila S, Georges A, Mishra K, Braund PS, d'Escamard V, Huang S, Margaritis M, Nelson CP, de Andrade M, Kadian-Dodov D, Welch CA, Mazurkiewicz S, Jeunemaitre X; DISCO Consortium; Wong CMY, Giannoulatou E, Sweeting M, Muller D, Wood A, McGrath-Cadell L, Fatkin D, Dunwoodie SL, Harvey R, Holloway C, Empana JP, Jouven X; CARDIoGRAMPlusC4D Study Group; Olin JW, Gulati R, Tweet MS, Hayes SN, Samani NJ, Graham RM, Motreff P, Bouatia-Naji N. Association of the PHACTR1/EDN1 Genetic Locus With Spontaneous Coronary Artery Dissection. J Am Coll Cardiol. 2019 Jan 8;73(1):58-66. doi: 10.1016/j.jacc.2018.09.085. PMID 30621952
- [Background] Turley TN, Theis JL, Sundsbak RS, Evans JM, O'Byrne MM, Gulati R, Tweet MS, Hayes SN, Olson TM. Rare Missense Variants in TLN1 Are Associated With Familial and Sporadic Spontaneous Coronary Artery Dissection. Circ Genom Precis Med. 2019 Apr;12(4):e002437. doi: 10.1161/CIRCGEN.118.002437. Epub 2019 Mar 19. PMID 30888838
- [Background] Turley TN, O'Byrne MM, Kosel ML, de Andrade M, Gulati R, Hayes SN, Tweet MS, Olson TM. Identification of Susceptibility Loci for Spontaneous Coronary Artery Dissection. JAMA Cardiol. 2020 Aug 1;5(8):929-938. doi: 10.1001/jamacardio.2020.0872. PMID 32374345
- [Background] Adlam D, Berrandou TE, Georges A, Nelson CP, Giannoulatou E, Henry J, Ma L, Blencowe M, Turley TN, Yang ML, Chopade S, Finan C, Braund PS, Sadeg-Sayoud I, Iismaa SE, Kosel ML, Zhou X, Hamby SE, Cheng J, Liu L, Tarr I, Muller DWM, d'Escamard V, King A, Brunham LR, Baranowska-Clarke AA, Debette S, Amouyel P, Olin JW, Patil S, Hesselson SE, Junday K, Kanoni S, Aragam KG, Butterworth AS; CARDIoGRAMPlusC4D; MEGASTROKE; International Stroke Genetics Consortium (ISGC) Intracranial Aneurysm Working Group; Tweet MS, Gulati R, Combaret N; DISCO register; Kadian-Dodov D, Kalman JM, Fatkin D, Hingorani AD, Saw J, Webb TR, Hayes SN, Yang X, Ganesh SK, Olson TM, Kovacic JC, Graham RM, Samani NJ, Bouatia-Naji N. Genome-wide association meta-analysis of spontaneous coronary artery dissection identifies risk variants and genes related to artery integrity and tissue-mediated coagulation. Nat Genet. 2023 Jun;55(6):964-972. doi: 10.1038/s41588-023-01410-1. Epub 2023 May 29. PMID 37248441
- [Background] Turley TN, Kosel ML, Bamlet WR, Gulati R, Hayes SN, Tweet MS, Olson TM. Susceptibility Locus for Pregnancy-Associated Spontaneous Coronary Artery Dissection. Circ Genom Precis Med. 2021 Aug;14(4):e003398. doi: 10.1161/CIRCGEN.121.003398. Epub 2021 Aug 13. No abstract available. PMID 34384238
- [Derived] Kok SN, Hayes SN, Cutrer FM, Raphael CE, Gulati R, Best PJM, Tweet MS. Prevalence and Clinical Factors of Migraine in Patients With Spontaneous Coronary Artery Dissection. J Am Heart Assoc. 2018 Dec 18;7(24):e010140. doi: 10.1161/JAHA.118.010140. PMID 30561271
- See also: Patient information on spontaneous coronary artery dissection — http://www.mayoclinic.org/diseases-conditions/spontaneous-coronary-artery-dissection/care-at-mayo-clinic/why-choose-mayo-clinic/con-20037794